CLINICAL TRIAL: NCT01051037
Title: Phase II Study Evaluating Safety and Efficacy of Stereotactic Body Radiotherapy and Radiofrequency Ablation for Medically Inoperable and Recurrent Lung Tumors Near Central Airways
Brief Title: Stereotactic Body Radiotherapy and Radiofrequency Ablation for Lung Tumors Near Central Airways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-08-026; 10-000656 (Other: UCLA/Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer
Keywords: lung tumors; central airways
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Subjects will undergo PET/CT simulation, 3 Fraction SBRT, RFA, and then undergo follow up.
  Interventions: Radiation: Stereotactic Body Radiation; Radiation: Radiofrequency Ablation

INTERVENTIONS:
Radiation: Stereotactic Body Radiation — 3 fraction of stereotactic body radiation therapy within 10 days.
  Other Names: SBR
Radiation: Radiofrequency Ablation — Subject will undergo radiofrequency ablation within 10 days of the last fraction of SBRT.
  Other Names: RFA

SUMMARY:
The purpose of this study is to demonstrate that combined stereotactic body radiotherapy and radiofrequency ablation is safe for patients with lung tumors near central airways.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary lung cancer, lung metastasis from another primary, or recurrent tumors in the setting of prior RFA or cryotherapy
* Tumors < 2 cm from trachea or zone of proximal bronchial tree (central tumors)
* Each tumor < 5 cm in size prior to treatment
* Medically inoperable patients as determined at the multidisciplinary thoracic tumor board, or medically operable patients who refuse surgery
* Criterion for medical inoperability include:

  * Overall clinical assessment at the UCLA thoracic tumor board
  * Reduced Pulmonary Function (FEV1, DLCO, etc) based on one major or two minor criterion as described below:
* Modified ACOSOG Criteria for medical inoperability:

  * Major Criteria: FEV1% < 50% or < 1L and DLCO < 50%
  * Minor Criteria: Age > 75, FEV1 51-60% predicted, or FEV1 1-1.2L, DLCO 51%-60% predicted, pulmonary hypertension, poor left ventricular function (EF < 40% or less), resting or exercise arterial pO2 < 55 mmHg, and pCO2 > 45 mmHg
* Age > 18 years old
* KPS > 70
* If a woman is of childbearing potential, a negative urine or serum pregnancy test must be documented.
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Prior thoracic radiation near the targets of interest
* More than 2 central tumor targets per patient
* Active infections requiring systemic antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-02-08 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Achieve at most of 20% subacute or chronic grade 3 or higher lng, cardiac, or upper GI toxicity rate in patients treated with SBRT/RFA. | 3 years

SECONDARY OUTCOMES:
Achieve no more than 15% decline from the pre-treatment pulmonary function parameter (FEV1, DLCO) post-SBRT/RFA. | 3 years
Achieve at least a 80% one-year local control (LC) rate by RECIST criterion or PET response (if applicable). | 3 years
Progression-free survival | 3 years
Overall survival | 3 years
Concentration of serum TGF-B as early biomarker for treatment-inducted normal tissue injury | 3 years
Concentration of serum VEGF as an early biomarker for response | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Percy Lee, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California, United States